CLINICAL TRIAL: NCT05112965
Title: An Open-Label, Multicenter Extension Study in Participants Previously Enrolled in a Genentech and/or F. Hoffmann-La Roche Ltd Sponsored Atezolizumab Study (IMbrella C)
Brief Title: An Extension Study in Participants Previously Enrolled in a Genentech and/or F. Hoffmann-La Roche Ltd Sponsored Atezolizumab Study (IMbrella C)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YO42713
Record Dates: First submitted 2021-11-02; First posted 2021-11-09 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — atezolizumab; Bevacizumab; Pemetrexed; Paclitaxel; enzalutamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Atezolizumab Monotherapy (Experimental): Participants will continue to receive atezolizumab monotherapy as per parent protocol, until disease progression or beyond if the participant continues to derive clinical benefit as judged by the investigator and if allowed by the parent study or local prescribing information until death; withdrawal of study consent; unacceptable toxicity; pregnancy; participant non-compliance; or study termination by the Sponsor, whichever occurs first.
  Interventions: Drug: Atezolizumab
- Combined Agents with Atezolizumab (Experimental): Participants will continue to receive atezolizumab with other agent(s) as per parent protocol, until disease progression or beyond if the participant continues to derive clinical benefit as judged by the investigator and if allowed by the parent study or local prescribing information until death; withdrawal of study consent; unacceptable toxicity; pregnancy; participant non-compliance; or study termination by the Sponsor, whichever occurs first.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Drug: Pemetrexed; Drug: Paclitaxel; Drug: Enzalutamide
- Comparator Treatment (Active Comparator): Participants will continue to receive comparator agent(s) as per parent protocol, until disease progression or beyond if the participant continues to derive clinical benefit as judged by the investigator and if allowed by the parent study or local prescribing information until death; withdrawal of study consent; unacceptable toxicity; pregnancy; participant non-compliance; or study termination by the Sponsor, whichever occurs first.
  Interventions: Drug: Bevacizumab; Drug: Pemetrexed; Drug: Paclitaxel; Drug: Enzalutamide

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered as a monotherapy or atezolizumab with other agent(s) as per parent protocol. Dosing regimen will continue in accordance with the parent study or at equivalent dose (if applicable) and at the same schedule as the parent study at the time of participant discontinuation from the parent study closure.
  Other Names: Tecentriq
  Arms: Atezolizumab Monotherapy; Combined Agents with Atezolizumab
Drug: Bevacizumab — Bevacizumab will be administered as directed per the parent study.
  Other Names: Avastin
  Arms: Combined Agents with Atezolizumab; Comparator Treatment
Drug: Pemetrexed — Pemetrexed will be administered as directed per the parent study.
  Arms: Combined Agents with Atezolizumab; Comparator Treatment
Drug: Paclitaxel — Paclitaxel will be administered as directed per the parent study.
  Arms: Combined Agents with Atezolizumab; Comparator Treatment
Drug: Enzalutamide — Enzalutamide will be administered as directed per the parent study.
  Other Names: Xtandi
  Arms: Combined Agents with Atezolizumab; Comparator Treatment

SUMMARY:
This is an open-label, multicenter, non-randomized extension study. Participants receiving atezolizumab monotherapy or atezolizumab combined with other agent(s) or comparator agent(s) in a Genentech or Roche-sponsored study (the parent study), who are eligible to continue treatment and do not have access to the study treatment locally, continue to receive study treatment in this extension study.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for continuing or crossing over to atezolizumab-based therapy at the time of rollover from the parent study, as per the parent study protocol, or
* Eligible for continuing the comparator agent(s) in a Genentech- or Roche-sponsored study as per the parent study protocol, with no access to commercially available comparator agent
* First dose of study treatment in this extension study will be received within 7 days of the treatment interruption window allowed by the parent study
* Continue to benefit from atezolizumab-based study treatment or from the comparator at the time of rollover from the parent study as assessed by the investigator
* Negative serum pregnancy test within 7 days prior to start of study treatment in women of childbearing potential
* For women of childbearing potential: agreement to remain abstinent or use contraceptive methods, and agreement to refrain from donating eggs
* For men: agreement to remain abstinent or use contraceptive measures, and agreement to refrain from donating sperm

Exclusion Criteria:

* Meet any of the study treatment discontinuation criteria specified in the parent study at the time of enrollment in the extension study
* Study treatment is commercially marketed in the patient's country for the patient-specific disease and is accessible to the patient
* Time between the last dose of treatment received in parent study and first dose in extension study is longer than the interruption period (±7 days) allowed in the parent study
* Treatment with any anti-cancer treatment (other than treatment permitted in the parent study) during the time between last treatment in the parent study and the first dose of study treatment in the extension study
* Permanent discontinuation of atezolizumab for any reason during the parent study or during the time between last treatment in the parent study and the first dose of study treatment in the extension study (if applicable)
* Any unresolved or irreversible toxicities during the parent study that required permanent discontinuation of study treatment, in accordance to the parent study or local prescribing information
* Ongoing serious adverse events that have not resolved to baseline level or Grade ≤1 from the parent study or during the time between the last treatment in the parent study and the first dose of study treatment in the extension study
* Any serious uncontrolled concomitant disease that would contraindicate the use of study treatment at the time of the extension study or that would place the patient at high risk for treatment-related complications
* Concurrent participation in any therapeutic clinical trial (other than the parent study)
* Pregnant or lactating, or intending to become pregnant during the extension study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Continued Access to Atezolizumab-based Therapy and/or Comparator Agent(s) | Up to approximately 4 years

SECONDARY OUTCOMES:
Percentage of Participants With Serious Adverse Events (SAEs) | Up to 90 days after the final dose of study treatment (up to approximately 4 years)
Percentage of Participants With Adverse Events of Special Interest (AESIs) | Up to 90 days after the final dose of study treatment (up to approximately 4 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (17):
- China (17):
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Union Hospital of Tongji Medical College, Dept. of Cancer Center, Wuhan, Hubei
  - Cancer Hospital of Shandong First Medical University, Jinan, Shandong
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - Beijing Cancer Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Changchun Cancer Hospital, Changchun
  - Jilin Cancer Hospital, Changchun
  - Hunan Cancer Hospital, Changsha
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Jiangsu Cancer Hospital, Nanjing
  - Shanghai Chest Hospital, Shanghai
  - Tianjin Cancer Hospital, Tianjin
  - The 2nd Hospital of Tianjin Medical University, Tianjin
  - Zhejiang Cancer Hospital, Zhejiang
  - Henan Cancer Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing